CLINICAL TRIAL: NCT03865719
Title: Ameliorate Childhood Obesity Risks From Newer Antipsychotics for Autism Spectrum Disorder
Brief Title: Weight Management Intervention for Youth and Young Adults With Autism Spectrum Disorder
Acronym: ACORN-ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Dana Rofey, Associate Professor of Psychiatry and Pediatrics, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY18120156
Record Dates: First submitted 2019-01-31; First posted 2019-03-07 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Autism Spectrum Disorder
Keywords: Second Generation Antipsychotics; Weight Management
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: An 11 session, 6 month healthy lifestyle program comprised of 30 to 45 minute sessions run by a dietician.
  Session 1 Getting Started/ anthropometric measures (weight, height, blood pressure and waist circumference)
  Session 2 Healthy Eating Habits/ anthropometric measures
  Session 3 Healthy Snacking Habits/anthropometric measures
  Session 4 Healthy Portions & Servings Habits/ anthropometric measures
  (BI-WEEKLY MEETINGS)
  Session 5 Healthy Shopping Habits/ anthropometric measures
  Session 6 Healthy Cooking & Mealtime Habits/ anthropometric measures .
  Session 7 Healthy Dining Out Habits/ anthropometric measures
  Session 8 Healthy Physical Activity Habits/ anthropometric measures
  (MONTHLY MEETINGS)
  Session 9 Healthy Eating Behavior Habits/ anthropometric measures
  Session 10 Healthy Problem Solving Habits/anthropometric measures
  Session 11 Maintaining a Healthy Lifestyle/ anthropometric measures
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Habits for Life Intervention (Other): Participants will receive the Healthy Habits for Life Intervention
  Interventions: Behavioral: Healthy Habits for Life

INTERVENTIONS:
Behavioral: Healthy Habits for Life — Healthy Habits for Life: 11-session, 6 month, one-on-one, dietician-lead weight management manualized treatment.

SUMMARY:
Psychotropic medications are the first-line treatment across several diagnostic categories encompassing severe mood disturbances and behavioral problems. The use of Second Generation Antipsychotics (SGAs) has increased in children with Autism Spectrum Disorder (ASD) in the last decade. However, SGAs are associated with serious metabolic side effects in youth that include cardiovascular disease, hypertension, and diabetes mellitus. This makes the public health impact of treating medication-induced metabolic disturbances almost as important as treating the mental illness itself. Improving health and reducing premature mortality in people with severe mental illness, the investigators propose to provide early weight management prevention, delivered by clinicians, for youth starting SGAs in order to target common modifiable health risk factors in the developmental process. This study will provide an urgently needed practical model for integrating weight management into academic- and community-based autism care.

DETAILED DESCRIPTION:
The innovations are four-fold: (1) adapting an evidence-based weight management treatment for youth/adolescents and young adults with Autism Spectrum Disorder (ASD); (2) training providers embedded within standard psychiatric care setting in an empirically-validated intervention for weight management; (3) utilizing a collaborative care model for weight management in psychiatric care for youth starting second generation antipsychotics (SGAs) to prevent/decelerate metabolic dysfunction; and (4) identifying factors that affect implementation into all Autism Treatment Network (ATN) sites. Given recent calls to move toward community-based obesity prevention approaches among high-risk youth, this study will provide an urgently needed intervention for adolescents and young adults with ASD on medications known to have untoward metabolic adverse effects. Moreover, this study will serve as a pilot mechanism to expand upon the findings in multiple ATN sites in a large-scale randomized control trial while measuring cardiometabolic outcomes. This pilot investigation has the potential to change standard of care within clinical practice that can be widely disseminated.

Aim 1: To refine the HH4L manual to meet the needs of youth/adolescents and young adults (IQ > 70) with ASD on SGAs by adding Cognitive Behavioral Therapy (CBT) techniques for managing behaviors related to eating and physical activity to an empirically-validated pediatric obesity manual and incorporating developmentally appropriate modifications for individuals with ASD with an emphasis on family-based changes.

Hypothesis 1.1: The CBT intervention will be feasible to deliver to adolescents and young adults with ASD and their family members.

Hypothesis 1.2: Participants will attend treatment regularly with low attrition (≤ 20%) and high attendance (>80%).

Aim 2: To test the efficacy of a psychiatrically-embedded weight management program for youth with ASD on SGAs. At the end of the 6-month program, youth receiving the weight management program (HH4L) will show improvements in:

Hypothesis 2.1: Maintained or decreased weight on BMI z-score (Primary Outcome)

Hypothesis 2.2: Ameliorated insulin resistance assessed by homeostatic model of assessment (HOMA-IR)(Secondary Outcome)

Hypothesis 2.3: Decreased systemic inflammation evaluated by circulating high sensitivity C-reactive protein (hs-CRP)

Exploratory Aim 3: To obtain a better understanding of how to support the effective implementation of HH4L into ATN sites.

Hypothesis 3.1. Identify organizational, clinician, and patient factors associated with effective implementation.

The main aim of this study is to adapt the Healthy Habits for Life manual to meet the needs of high-functioning adolescents and young adults with ASD who gain >7% of initial body weight while taking a SGA (or >5% if overweight/obese). HH4L is a CBT, MI, and family-based weight management intervention. However, proposed changes may include emphasizing the effects of SGAs on appetite, adapting cognitive foci to behavioral, emphasizing the role of family in stimulus control, and focusing on sneak eating.

HH4L-ASD will involve eleven 45-minutes sessions over a 6-month period. Dependent measures will include physiological outcomes (e.g., Body Mass Index; BMI) and emotional/behavioral outcomes (e.g., Aberrant Behavior Checklist) collected at baseline and monthly there-after. While outcome data will inform next steps, the main aim of this pilot is to create a manual that can be implemented at all ATN sites.

Study Flow: Families will be informed of the study by staff at the Pitt ATN. Interested families will undergo either a telephone or face-to-face screen, at which time they will be provided with additional information regarding study aims and expectations. At a subsequent in-person screen/baseline assessment, the child/family will have all questions answered and will sign an informed assent and consent. All participants will receive treatment. There are 4 weekly sessions, 4 bi-weekly sessions, and 3 monthly booster sessions over a 6 month period. Given that some families come from far away and there are often barriers that impact patient attendance, 25% of all sessions will be permitted to be via phone or text sessions. These are options in line with prior investigations by PI Rofey. These telehealth standards are similar to the research group's prior work validating the effectiveness of HH4L. Participants will work one-on-one with a practitioner who has been delivering HH4L for over a decade. Retention rates are expected to be commensurate with similar studies (~ 90%).

Data Management. The Principal investigators (PIs) will oversee all aspects of data management. With the consultation of the Massachusetts General Hospital Data Coordinating Center (DCC), the PIs and coordinator will develop an operations manual to standardize all procedures and staff training. All study participants will be assigned unique study identifiers that will appear on all data collection instruments, tapes, documents, and files used in the statistical analysis and manuscript preparation. The DCC also has specific data quality measures that will be implemented.

Statistical Analyses Data will be summarized using sample means or proportions along with 95% confidence intervals within each study arm.

Attrition and Missing Data. Every effort will be made to minimize the amount of attrition and missing data. The current research group has a history of successful retention of subjects in clinical research protocols. Participants are able to conveniently schedule research visits to correspond with regularly scheduled clinical appointments. Retention rates in 2 similar random control trials range from 80-90%. Follow-up assessments will be attempted even if a participant has dropped out of the training program. The investigators will also offer shortened assessments to convert initial refusals.

Sample size. The sample size (25 participants) is based on feasibility considerations for the recruitment period. With 25 participants enrolled, the exact 95% confidence interval on a completion rate of 80% is 59.30%-93.17%. Assuming 80% have a 6-month BMI measurement, and 80% are lower than at baseline, the exact 95% confidence

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Autism Spectrum Disorder based on Autism Diagnostic Observation Schedule, Second Edition (ADOS-2) and The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria.
2. Clinically stable on current SGA treatment regimen with olanzapine, quetiapine, risperidone, aripiprazole, ziprasidone, or clozapine.
3. The patient meets one of the following criteria:

   If the participant is under 20 years old, the participant either:
   1. has a BMI greater than or equal to 85th percentile, corrected for age and sex, AND has a documented 3% increase or greater in BMI within the last 12 months, while on SGAs, or
   2. has persistent and unrelenting BMI percentile at or above 98%, corrected for age and sex (3% change in BMI is not necessary).

   If the participant is 20 years old or older, the participant either:
   1. has a BMI greater than or equal to 30 AND has a documented 3% increase or greater in BMI within the last 12 months, while on SGAs, or
   2. has persistent and unrelenting BMI at or above 40 (3% change in BMI is not necessary)4. Involvement of at least one parent or guardian if ≤ 18 years of age. If > 18, an adult caregiver living with the participant must agree to complete the parent/guardian measures.
4. Age between 8 and 26, inclusive.
5. Prior to the study, minor participants must provide assent to participate in the study, and their parents (guardians) must provide written informed consent. Individuals > 18 will provide written consent.

Exclusion Criteria:

1. IQ < 70.
2. Recent suicide attempt (within 1 month of study entry) or illness severity requiring acute psychiatric hospitalization within 30 days of study entry.
3. Current weight management treatment with CBT by an appropriately trained provider using a manual. If currently receiving treatment, willingness to suspend treatment for 12-week acute treatment phase of study.
4. New mood stabilizer, selective serotonin reuptake inhibitor (SRRI) or stimulant medication. If patient has been stable on psychotropic medication for 30 days, inclusion is permitted.
5. Pregnant.
6. Diagnosis of diabetes.
7. Participant and/or parent/caregiver/service provider/partner/friend of the participant unwilling or not able to commute for study visits
8. Unwilling to have bloodwork.
9. Taking medications that affect bodyweight, other than SGAs, for less than a month (e.g., Metformin, Prednisone, Topiramate, or any other medications, in the opinion of the Site Principal Investigator, would deem as a medication that would affect bodyweight).

Ages: 8 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) z-score | Change from Baseline to intervention completion at 6 months
  BMI z-scores will be calculated from participant height(cm), weight(kg), sex and age
Inflammation as indicated by change in circulating high sensitivity C-reactive protein (hs-CRP) | Change from Baseline to intervention completion at 6 months
  hs-CRP level from blood work completed at local lab

SECONDARY OUTCOMES:
Implementation effectiveness | Month 6
  Parent/Caregiver and Research team completed questionnaire regarding project implementation. There are 12 items to be rated on Likert scales as well as 3 open-ended questions. There are no scales associated with this survey. The results will help us draw a qualitative picture of the parent satisfaction with the program and research team appraisal of the effectiveness of the program across subjects.
Change in Waist circumference | Change from Baseline to intervention completion at 6 months
  Waist circumference measured in centimeters by dietician will be measured in duplicate, midway between the lowest rib and the superior border of the iliac crest, with a flexible tape.
Change in Blood pressure | Change from Baseline to intervention completion at 6 months
  Blood pressure measured in millimeters of mercury (mmHg) by dietician using a portable blood pressure cuff at intervention appointment
Change in Lipid Panel Lab Values | Change from Baseline to intervention completion at 6 months
  Fasting Lipids Panel from blood work completed at local lab (in mg/dL): Cholesterol, HDL, Cholesterol/HDL Ratio (calculated), LDL, Triglycerides
Change in Glucose Serum | Change from Baseline to intervention completion at 6 months
  Glucose serum level from blood work completed at local lab, mg/dL
Change in Insulin | change from Baseline to intervention completion at 6 months
  Insulin level from blood work completed at local lab, µIU/mL
Change in HOMA-IR | change from Baseline to intervention completion at 6 months
  HOMA-IR is a method used to quantify insulin resistance (fasting glucose X fasting insulin / 22.5).
Change in aberrant behaviors | change from Baseline to intervention completion at 6 months
  Change in aberrant behaviors as measured by the Aberrant Behavior Checklist (ABC). The ABC is comprised of 58 items aimed to capture specific behavioral symptom areas: Irritability (15 items), Lethargy (16 items), Sterotypy (7 items), Hyperactive/Noncompliace (16 items)/Inappropriate Speech (4 items).
  To score the ABC, the individual items for each subscale are simply summed to their respective subtotals with higher scores reflective of more pervasive symptoms on that subscale.
Change in emotional dysregulation | change from Baseline to intervention completion at 6 months
  Change in emotional dysregulation as measured by the Emotion Dysregulation Inventory with 30 items on two factors: (1) Reactivity, characterized by intense, rapidly escalating, sustained, and poorly modulated negative emotional reactions, and (2) Dysphoria, characterized by anhedonia, sadness, and nervousness. Items are rated on the following scale to reflect current behavior: and how much of a problem it has this been in the preceding 7 days?:
  Not at all (0, never happens) Mild (1, Present occasionally) and/or does not cause too much of a problem Moderate (2, Happens less than half the time and/or causes some problems Severe (3, Happens at least half of the time and/or substantially interferes Very Severe: 4, Almost always happens and/or causes a serious problems
  Scores for items on each factor are summed for a total scale score. Higher scores suggest more emotional dysregulation on that specific factor.
Change in parenting stress | change from Baseline to intervention completion at 6 months
  Change in participant's parent's/caregiver's stress as measured by the Parenting Stress Short Form (PSI-SF), a 36 items assessing Total Stress is calculated by summing the raw score from three scales: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child. A higher score represents higher parent stress.
Change in weight loss behaviors | change from Baseline to intervention completion at 6 months
  Change in weight loss behaviors as measured by the Weight Loss Behavior Stage of Change Scale (WLB_SOC). The numerical values on the WLB-SOC questionnaire directly correspond to the five Stages of Change:1 = pre-contemplation; 2 = contemplation; 3 = preparation; 4 = action; 5 = maintenance The questionnaire has 5 sections: Potions, Dietary Fat, Fruits, Vegetables, Usual Physical Activity. For sections that have 9 or 10 questions (i.e., Portions, Fruits and Vegetables, Usual Physical Activity), the SOC is determined by using the third lowest stage for the behavioral items. For sections that have 11 questions (Dietary Fat), the SOC is determined by using the fourth lowest stage indicated for the behavioral items. Items answered "N/A" or left blank are scored as a "1".
Change in physical activity habits | change from Baseline to intervention completion at 6 months
  Change in physical activity habits as measured by the Modifiable Activity Questionnaire (MAQ). This measure is a self-reported questionnaire that records frequency and duration of different levels of physical activity. The MAQ assesses current physical activity during both work and leisure time, as well as some inactivity. The hours per week of all activities are summed to determine total hours per week.

CONTACTS AND LOCATIONS:
Overall Officials: Dana L Rofey, PhD, Principal Investigator — University of Pittsburgh; Benjamin L Handen, PhD, BCBA-D, Principal Investigator — University of Pittsburgh
Locations (1):
- Autism Treatment Network Site at Merck Child and Adolescent Outpatient Clinic, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No